CLINICAL TRIAL: NCT03444116
Title: Long-Term Outcomes of Femoral Derotation Osteotomy for Individuals With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Tom F Novacheck, Pediatric Orthopedic Surgeon, Gillette Children's Specialty Healthcare
Other Study IDs: Study 00000239
Record Dates: First submitted 2018-02-07; First posted 2018-02-23 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy; Femoral Derotation Osteotomy; Outcomes
MeSH Terms: conditions — Cerebral Palsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (+FDO): Patients who underwent an FDO
  Interventions: Diagnostic Test: Motion Analysis; Diagnostic Test: sterEOS Imaging of Lower Extremities; Behavioral: Surveys
- Controls (-FDO): Same as cases but did not undergo an FDO
  Interventions: Diagnostic Test: Motion Analysis; Diagnostic Test: sterEOS Imaging of Lower Extremities; Behavioral: Surveys

INTERVENTIONS:
Diagnostic Test: Motion Analysis — Gait and Motion Analysis, comprised of 3-dimensional kinematics and kinetics, electromyography, energy expenditure, and physical exam (range of motion, strength, spasticity, etc.)
Diagnostic Test: sterEOS Imaging of Lower Extremities — Bi-planar imaging of the lower extremities to evaluate femoral anteversion and hip dysplasia and subluxation.
Behavioral: Surveys — 9 surveys assessing function, activity, participation, pain, quality of life, and treatment history.

SUMMARY:
Excessive anteversion is commonly observed in the cerebral palsy (CP) population. This can be treated by an orthopedic surgery, called femoral derotation osteotomy (FDO), to de-rotate the femur. It is a vital aspect of patient care to understand if the effects of an FDO are maintained long-term. The results of this study will have direct clinical impact by equipping providers with the necessary information to counsel families by providing families the information needed to make the most informed decision possible about this aspect of their child's healthcare.

DETAILED DESCRIPTION:
Excessive anteversion is commonly observed in the CP population. If individuals do not internally rotate their femurs as a compensation for this bony torsion, excessive anteversion decreases the coronal plane moment arm of the hip abductors-a phenomenon often called lever arm dysfunction. Considering that adequate hip abductor strength is a crucial factor for normal walking and many other functional activities, the compensatory mechanism theory hypothesizes that individuals with excessive anteversion will internally rotate their hips to restore the coronal plane moment arms. Excessive internal hip rotation (IHR) is observed in the gait of approximately 50% of individuals with CP. It has been postulated, though, that while IHR may restore hip abductor function, it is cosmetically unappealing and may lead to trips and falls. Therefore, FDOs are considered the standard treatment for correcting excessive anteversion and IHR in individuals with CP. Notably, it is one of the top two orthopedic surgeries performed at Gillette Children's Specialty Healthcare. Among the ~4000 individuals with CP who have been seen in the gait lab, almost 1350 individuals (>2200 limbs) have undergone at least one FDO.

Short-term (~12 months postoperative) improvements of transverse plane hip rotation during gait range from only 33% to 94%. Despite FDO's widespread use, long-term outcomes of the procedure have only begun to be studied, with our 2016 study the only one that included a control group. Without a control group, the natural history of bony remodeling or gait adaptations is unknown. However, our prior study is limited by two main factors, 1) all data were extracted from our database retrospectively, so the potential for a large bias exists since outcomes reflect only patients with clinically-initiated gait visits, and 2) outcomes of hip abductor function were only measured by hip rotation (or hip abductor moment during gait, which is only available for individuals who can walk without assistive devices), so the true ability of the hip abductors to generate moment has not been tested. Furthermore, the vast majority of individuals were <18 years old at their "long-term" visit (~5 years after their preoperative gait visit), which precedes the reported gait or functional decline more commonly occurring in one's 20s and beyond.

Counseling families on the long-term outcomes after an FDO is currently not possible and is necessary for families and health-care providers to make informed decisions. It remains unclear whether individuals who receive an FDO experience long-term beneficial effects on function, activity, and comfort as compared to those who receive other or no treatment for their excessive anteversion and/or IHR.

Briefly, anteversion as measured by the trochanteric prominence angle test (TPAT) is the most common method used by clinicians to determine if an FDO is warranted, in addition to anteversion being an important predictor of predicted short-term outcomes after an FDO23. However, data from our lab suggests that there is 10-15° of measurement error associated with this method. As such, our secondary purpose was to compare anteversion as measured by the TPAT to that of a radiographical gold standard, EOS. EOS delivers 4-30 times less radiation to the gonads and lower extremities compared to computed tomography (CT)24, making it very suitable for research purposes. Additionally, accuracy of quantifying femoral anteversion is not compromised versus the current gold standard, CT, with a mean difference of ~3° reported.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral CP (i.e., hemiplegics excluded)
* Minimum age of 25 years presently
* Had a preoperative gait analysis
* Underwent only 1 external, proximal FDO per side
* Minimum 5 years since an FDO
* FDO implants have been removed
* No prior pelvic osteotomy
* Able to speak and read English
* Not pregnant

Control group (-FDO):

* Same as cases, except no FDO
* Matched to cases at baseline (using a matching algorithm)

Exclusion Criteria:

* none

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former/current patients at Gillette Children's Specialty Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Gait and Motion Analysis | long-term research visit (on average, ~10 years post-baseline)
  Compare gait kinematics and kinetics across groups
sterEOS imaging | long-term research visit (on average, ~10 years post-baseline)
  femoral anteversion determined by 3-D reconstruction of bi-planar sterEOS imaging
Change in Gait and Motion Analysis | baseline (qualifying exam, pre-FDO or gait analysis at which controls matched cases) compared to long-term research visit (on average, ~10 years post-baseline)
  Compare change in gait kinematics and kinetics within groups

SECONDARY OUTCOMES:
sterEOS imaging | long-term research visit (on average, ~10 years post-baseline)
  Assess hip dysplasia and/or subluxation in qualifying limb across groups
Number of hip abduction repetitions | long-term research visit (on average, ~10 years post-baseline)
  Assess hip function across groups
Seconds to complete Timed Up and Go | long-term research visit (on average, ~10 years post-baseline)
  Assess function across groups
Quality of Life as assessed by WHOQOL-bref | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Pain as assessed by the Brief Pain Inventory | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Fear of Falling as assessed by Falls Efficacy Scale-International | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Hip Function as assessed by Harris Hip Function | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
General Function as assessed by Functional Assessment Questionnaire | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Walking Function as assessed by Function Mobility Scale | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Participation as assessed by Child/Adolescent Frequency of Participation Questionnaire | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey
Satisfaction with Life as assessed by Deiner Satisfaction with Life Scale | compare scores across groups at long-term research visit (on average, ~10 years post-baseline)
  self-reported survey

CONTACTS AND LOCATIONS:
Overall Officials: Tom F Novacheck, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No